CLINICAL TRIAL: NCT05283668
Title: The Adjunctive Effect of Injectable Platelet Rich Fibrin on Healing and Patient Satisfaction Following Laser Gingival Depigmentation (A Randomized Clinical Trial With Histological Analysis)
Brief Title: Effect of Injectable Platelet Rich Fibrin on Healing and Patient Satisfaction Following Laser Gingival Depigmentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ola Mohamed Ezzatt, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FD-ASU -2021
Record Dates: First submitted 2022-02-28; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Gingival Pigmentation
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (LASER WITH I-PRF) (Experimental): Eight sites that were treated with laser method for gingival depigmentation, followed by intra-mucosal field injection of I-PRF
  Interventions: Biological: i-PRF; Procedure: Diode Laser
- (LASER WITHOUT I-PRF) (Active Comparator): Eight sites that were treated with laser technique for gingival depigmentation only
  Interventions: Procedure: Diode Laser

INTERVENTIONS:
Biological: i-PRF — * Local anesthesia was achieved using field block technique.
  * A soft tissue diode surgical laser unit was used in a contact method using a flexible fiber optic hand piece with initiated tip.
  * Laser irradiation parameters were adjusted as follows: Wavelength [940 ± 10 nm], irradiation mode [contact continuous wave], Power [2 W] and 300 μm fiber tip diameter (Jokar et al., 2019).
  * The treatment was depigmentation by laser thin injection by I-PRF Post-operative instructions Instruct the patients to avoid tooth brushing on the day of surgical treatment to prevent mechanical trauma and allow re-epithelialization.
  Arms: (LASER WITH I-PRF)
Procedure: Diode Laser — Local anesthesia was achieved using field block technique.
  * A soft tissue diode surgical laser unit was used in a contact method using a flexible fiber optic hand piece with initiated tip.
  * Laser irradiation parameters were adjusted as follows: Wavelength [940 ± 10 nm], irradiation mode [contact continuous wave], Power [2 W] and 300 μm fiber tip diameter (Jokar et al., 2019).
  Post-operative instructions Instruct the patients to avoid tooth brushing on the day of surgical treatment to prevent mechanical trauma and allow re-epithelialization.

SUMMARY:
The objectives of the present study are to:

1. Evaluate the effect of I-PRF injection following laser gingival depigmentation technique on the healing period as a primary objective.
2. Assess patient satisfaction following the procedure in terms of pain and esthetic outcome as a secondary objective.

DETAILED DESCRIPTION:
Dental esthetic needs are increasing in recent years with a greater demand on pleasant appearance; including a healthy set of dentitions but also esthetically improved gingival appearance, especially when it is located in the anterior labial region. Physiologic gingival hyperpigmentation affects numerous people of different ethnic backgrounds.

Gingival depigmentation is defined as a periodontal plastic surgical procedure that are aimed at removing the pigmented gingiva and methods aimed at masking the pigmented gingiva. Techniques of gingival depigmentation can be classified as; chemical methods mainly by ascorbic acids, surgical methods, electrosurgery, cryosurgery, radiosurgery, and lasers.

The study was conducted on eight patients seeking treatment for their gingival hyperpigmentation for esthetic reasons. A total number of 16 sites of facial gingival hyperpigmentation were treated, two in each patient in a split mouth technique.

* Group I (LASER with I-PRF): Included eight sites that were treated with laser technique for gingival depigmentation, followed by intramucosal field injection of I-PRF (as study group).
* Group II (LASER): Included eight sites that were treated with laser technique for gingival depigmentation (as a control group).

The clinical outcomes were assessed for each patient: at baseline (pre-operative), post-operative, one week, one month. Clinical assessment was done by measuring DOPI, clinical wound healing, VAS and patient satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Male and female with age range from 16 to 45 years old.
* Systemically free from any disease as evidenced by the health questionnaire guided by modified Cornell medical index (Pendleton et al., 2004).
* Gingival hyperpigmentation on maxillary and mandibular labial keratinized gingiva score 3 (Dummett et al., 1964).
* Patient with thick gingival phenotype (>1.5mm) (Claffey and Shanley, 1986).

Exclusion Criteria

* Pregnant and lactating women.
* Smokers.
* Gingival pigmentation associated with occupational Hazards.
* Patients with missing anterior teeth.
* Patients with any metallic restoration related to anterior teeth or undergoing orthodontic treatment.
* Vulnerable groups (prisoners, handicapped and orphans).

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Dummet oral pigmentation index | 1 month
  the degree of gingival pigmentation will be scored as: 0 = pink tissue [no clinical pigmentation]; 1 = mild light brown tissue [mild clinical pigmentation]; 2 = medium brown or mixed brown and pink tissue [moderate clinical pigmentation]; or 3 = deep brown/ blue-black tissue [heavy clinical pigmentation]
Clinical wound healing | 1 week
  scored as follows:
  1) Complete reepithelialization, 2) Incomplete reepithelialization, 3) ulcer and 4) tissue defect or necrosis

SECONDARY OUTCOMES:
Satisfaction questionnaire | 1month
  score the degree of satisfaction about cosmetic outcomes of treatment
Visual analogue scale (VAS) score for pain assessment | 1month
  Pain assessment will be performed using a 10-cm (100 mm) horizontal continuous scale marked "no pain" on the left and "maximum pain" on the right side of the scale. The scores were as follows: no pain (0), slight pain (0.1-3.0 mm), moderate pain (3.1-6.0 mm), and severe pain (6.1-10 mm)
Histological assessment | 1 week
  The mean of epithelial thickness for each case was calculated

CONTACTS AND LOCATIONS:
Overall Officials: Ola Ezzatt, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Available on request at principle investigator

REFERENCES:
- [Derived] Ibrahim SSA, Mandil IA, Ezzatt OM. Injectable platelet rich fibrin effect on laser depigmented gingiva: a clinical randomized controlled split mouth trial with histological assessment. J Appl Oral Sci. 2024 Mar 25;32:e20230307. doi: 10.1590/1678-7757-2022-0307. eCollection 2024. PMID 38536994